CLINICAL TRIAL: NCT06711354
Title: B-cell Depletion in Offspring to Women With MS and Rituximab Treatment Before or During Pregnancy
Brief Title: B-cell Depletion in Offspring to Women With MS Under Immunomodulatory Treatment
Status: Not yet recruiting | Type: Observational
Sponsor: Region Stockholm (Other Government)
Collaborators: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 142682
Record Dates: First submitted 2024-11-26; First posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-05

CONDITIONS: Multiple Sclerosis; B-Cell Deficiency; Offspring, Adult; Immunosuppression; Pregnancy Related
MeSH Terms: conditions — Multiple Sclerosis | interventions — Rituximab; ocrelizumab; ofatumumab

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — Venous blood samples from mother analyzing immunoglobulin levels and B-cell levels as part of clinical routine. Additional analysis of anti-CD20 medication concentration as part of present study.
  Capillary blood samples from child analyzing antibodies produced through vaccination or infection.
  Dry blood spot from existing blood samples from child, obtained during routine screening, with complementary analysis of CD19, KREC and anti-CD20 medication concentration.
  Breast milk analysis of anti-CD20 medication concentration.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Mother exposed to anti-CD20 ab: Mothers with MS exposed to monoclonal anti-CD20 antibody (Rituximab 500 mg iv alternatively Ofatumumab 20 mg sc or Ocrelizumab 300-600 mg iv) within 12 months before pregnancy or during pregnancy.
  Interventions: Drug: Anti-CD20 Monoclonal Antibody
- Mother exposed to other DMT: Mothers with MS exposed to disease modifying therapy other than Rituximab, Ofatumumab or Ocrelizumab within 6 months before pregnancy
- Mother without DMT exposure: Mothers with MS without exposure to disease modifying therapy within 6 months before pregnancy

INTERVENTIONS:
Drug: Anti-CD20 Monoclonal Antibody — Injection of monoclonal anti-CD20 antibody as immunomodulatory treatment of multiple sclerosis
  Other Names: Rituximab; Ocrelizumab; Ofatumumab
  Groups: Mother exposed to anti-CD20 ab

SUMMARY:
The overall aim of the study is to gain knowledge about consequences for the child´s humoral immunosystem in mothers with multiple sclerosis and due to their immunomodulating treatments. Of special interest is when the mother is treated with monoclonal CD20-antibody like rituximab, ocrelizumab and ofatumumab shortly before (within six months prior to conception) and during pregnancy. Specific aims of the study are to:

* Investigate if the humoral immunosystem is fully functioning at birth in children born to mothers with MS
* Investigate if the humoral immunosystem at birth in children born to mothers with MS is influenced by the mothers immunomodulating treatment
* Investigate if monoclonal CD20-antibodies are fully eliminated in women treated with monoclonal CD20-antibodies within 12 months prior to conception.
* Determine if children who have been exposed to monoclonal CD20-antibody in utero have reduced markers of successful B-cell production at birth.
* Investigate the response to the Rota virus vaccine, a life-vaccine that is offered 6 weeks after birth to all children born after September 2019, in children to women treated with rituximab before or during pregnancy.
* Investigate the response to other vaccines (DTP, Polio, HiB, pneumococcus given at 3 and 5 months after birth) the earliest one months after vaccination.
* Investigate the occurrence of infections in the first-year post-partum for the mother and child due to hypogammaglobulinemia, b-cell depletion, and exposure to monoclonal CD20-antibody.
* Investigate if oral exposure to rituximab through mother´s breastmilk is resulting in B-cell reduction in the child.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a chronic inflammatory disorder of the central nervous system affecting more women than men and typically manifests during reproductive ages (1). The disease and associated treatments therefore have a large impact on family planning. While trying to conceive most clinicians recommend discontinuation of disease-modifying drug use (DMD) before conception unless the risk of disease worsening outweighs the risk to the fetus (2,3). Patients with active disease may need to continue DMD treatment until conception or even during pregnancy. Furthermore, given that nearly half of all pregnancies are unplanned (4-6) women with MS may occasionally become pregnant during or shortly after receiving treatment. As such, gathering information on the effect of pregnancy exposure to DMD is crucial for the management of reproductive issues in women with MS.

Rituximab, a chimeric monoclonal B cell-depleting anti-CD20 antibody, is frequently used off-label for the treatment of MS in Sweden (7). The drug targets CD20 on the cell surface of B cells and effectively depletes them. Previously recommendations of rituximab was withdrawn at least one year prior to a planned pregnancy. Given the pharmacokinetics with a halftime of around 24 days current Swedish guidelines accept a minimum of 3-4 months between last infusion and conception. Rituximab is a chimeric antibody of the immunoglobulin G1 kappa type and is therefore actively transported over the blood-placenta barrier, mainly during the third trimester but starting already in the second trimester. Small case series and reports show that rituximab administered during the third trimester suppresses neonatal b-cell development (8-12). After six months, usually, b-cells levels normalize but effects may not be clinically apparent at birth but may influence response to vaccinations early in life and increase susceptibility to infections.

Severe combined immunodeficiency (SCID) is included in the Swedish national neonatal disease screening program, testing is performed at Centrum för Medfödda Metabola Sjukdomar (CMMS), in parallel with screening tests for other diseases, on blood samples in the form of dry blood spots (DBS) taken within 48 hours after birth. The SCID screening consists of assessing markers of T and B cell production, T-cell receptor excision circles (TREC) (13) and kappa-deleting recombination excision circles (KREC)(14) , respectively. Both are circular fragments of DNA that are excised during the gene rearrangements necessary for the formation of functional T- and B-cell receptors. KRECs are formed during the rearrangement of the kappa light chain gene and occurs in the bone marrow at the small pre-B-cell stage. CD20 is already expressed on the surface of these B-cell precursors and they may therefore be targeted by rituximab and other monoclonal anti-CD20 antibodies (15). Each cell forms one KREC copy, which by necessity is passed to only one of the cells after cell division. Consequently, a proportion of mature B-cells in the circulation will also carry KRECs, and because they express CD20 they may be depleted by rituximab.

We hypothesize that if rituximab inhibits B-cell formation in the fetus of a pregnant mother treated with the drug, this can be detected in the form of reduced KREC results. A case report that describes a child of a rituximab treated mother that had reduced KREC results at birth has been published suggesting that such effects occur (16). It has also been shown that broad immunosuppressants, in particular the purine analogue azathioprine, cause some KREC results that are under the cutoff in the neonatal screening in Sweden (17). More knowledge is needed regarding the safety of rituximab for the fetus during pregnancy to facilitate clinical decisions in this complex situation, being able to identify offspring with insufficient B-cell counts and consequently at higher risks for infection and influence of vaccination responds. Such knowledge will facilitate clinical decisions and may help identify offspring with insufficient B cell counts and consequently at higher risks for infection and poor vaccine response.

The experimental plan includes a retrospective part as well as a prospective part.

The retrospective part of the study will take advantage of already existing blood samples from the national newborn screening program and examine the KREC results of all children born to rituximab treated mothers with MS in Stockholm during the past 10 years. Information on DMD treatment, time of conception, B-cell level, immunoglobulin levels in the mothers at the end of each trimester are routinely collected and recorded in the Swedish Multiple Sclerosis registry (SMSreg). Mothers that have been treated with monoclonal CD-20 antibodies and other MS specific DMTs during pregnancy or within twelve months before conception and have successfully delivered a child will be included in the study. After informed consent has been received from the parents our collaborators at CMMS will extract KREC results if available from either the screening program or the preceding pilot study(17). If results are not available, the DBS samples will be retrieved and KREC analyzed specifically for this study. If the combined KREC results are ambiguous we have the option to retrieve DBS samples for all included children and perform an in-house assay developed at CMMS to confirm B-cell deficiency by determining abundance of CD19 transcripts in the sample. Furthermore, to be able to correlate B-cell deficiency to drug concentration in the child, DBS can be sent for drug level detection to our collaborators at the Haukeland University Hospital laboratory. The mothers B-cell deficiency and its consequence on immunoglobulin levels will also be assessed in the analysis.

In the prospective part of the study we plan to address if a reduction in the levels of KREC and/or CD19+ B-cells at birth of offspring to women with MS has clinical significance. Mothers with MS, regardless of treatment, that have successfully delivered or will deliver a child will be asked for informed consent included if applicable.

1. At clinical routine venous blood sampling immunoglobulin and B-cell levels are obtained. Additional samples, during clinical routine visit, in the becoming mother will allow analysis of drug concentration at the end of every trimester and 3 months post partum.
2. Within 1-12 months postpartum and after vaccination capillary blood samples from the child will be analyzed to detect antibodies induced by vaccination or infections to secure the ability to be able to develop antibodies despite being exposed to monoclonal CD20-antibodies in-utero or via breastmilk.
3. PKU-test is taken in the child within routine but additional analysis on drug levels and KREC will be analyzed as well as determining abundance of CD19 transcripts.
4. Within our routine contacts with the MS patient (mother) we will ask for infections in both, the mother and the child at 3 months and 1 year post-partum.

After informed consent has been received from the parents our collaborators at CMMS will also extract KREC results if available from the screening program. If results are not available, the DBS samples will be retrieved and KREC analyzed specifically for this study. If the combined KREC results are ambiguous we have the option to retrieve DBS samples for all included children and perform an in-house assay developed at CMMS to confirm B-cell deficiency by determining abundance of CD19 transcripts in the sample.

Primarily Rota virus vaccine will be considered because it is the earliest vaccination in the national vaccination program, offered at 6 weeks of age. Antibody levels for other vaccines or infections may be tested if deemed relevant. A detailed infectious and general medical history via the parents will be obtained at routine contacts between patient and health care and comparison of adverse outcomes between children with mothers exposed to rituximab and children to mothers with MS but without rituximab treatment within 12 months prior to conception as well as for children with and without apparent reduction in the levels of KREC and/or B-cell depletion due to in utero exposure to rituximab and children with normal KREC levels will be summarized.

In Canada, Germany and the US, breastfeeding despite receiving anti-CD20 antibody therapy is getting more common, assuming the antibody cannot be enterally absorbed hence eliminated fecally ungraded. Swedish recommendations at present are cessation of breastfeeding when starting DMT however more women choose to breastfeed regardless. We would like to offer a follow-up with breastmilk samples and blood samples in the child one month after drug application for drug level detection in breastmilk and child and B-cell level analysis in the child.

Sample analysis of B-cell levels, IgG and IgM levels as well as specific antibodies as detection for immune responds to vaccination will be analyzed with clinically established methods via the lab at Karolinska University Hospital and Lennart Svenssons lab in Linköping, Sweden. Blood sampling from the child will be performed at specialized blood sampling centers for children e.g. Karolinska university hospital. KRECs and abundance of CD19 transcripts will we analyzed in dried blood spots at CMMS with an established method within the clinics. As there is no existing established high-quality method in Sweden, we will have to send drug level analysis to the Bergen University in Norway, our collaborator. They will use ELISA and high-performance liquid chromatography-electrospray ionization mass spectrometry method to analyses drug levels in blood, breast milk and dried blood spots.

Descriptive data and differences in drug levels, cell levels, infection rate and KREC levels between women with MS who have been exposed to ant-CD20 antibodies and not close to their pregnancy and their offspring will be tested with chi2-tests or Wilcoxon rank sum test, where appropriate. IgG levels will be analyzed using a linear mixed effect model, including number of doses of administered DMT (i.e. RTX or other DMTs) as random effect, while age, sex, previous DMT, administered DMT and the interaction of doses and administered DMT as fixed effects. P-values <0.05 will be considered statistically significant. Non-parametric variables will be presented as median (range), and normally distributed variables as mean (SD).

The dilemma of balancing the mothers need for effective treatment against potential harmful effects to the fetus is a common clinical problem. It is virtually impossible to study the effects of drugs on the developing child apart from gathering observational data from individual cases where, for any reason, the mother did receive a certain drug. In Sweden the conditions are especially good to gather information on the effects of in utero exposure to B-cell depleting drugs because the unique propensity to treat MS-patients with monoclonal CD20-antibodies (e.g. rituximab) in combination with a newborn screening program that includes a marker for B-cell deficiency. The study results will have direct impact on the clinical management of MS-patients with aggressive disease and family planning wishes.

ELIGIBILITY:
Inclusion Criteria:

* Definite diagnosis of multiple sclerosis in mother AND
* Administration of Rituximab, Ocrelizumab or Ofatumumab within 12 months or during established pregnancy OR
* Administration of other immunomodulatory treatment within 12 months or during established pregnancy OR
* No administration of immunomodulatory treatment within 12 months or during established pregnancy

Exclusion Criteria:

* Treatment with stem cell transfusion

Max Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Women with definite diagnosis of multiple sclerosis who are pregnant are divided in study groups based on treatment 12 months prior to pregnancy. Study groups consist of treatment with monoclonal anti-CD20 antibodies, other immunomodulatory treatment and absence of immunomodulatory treatment respectively.
  Population also consist of offspring to women as described above with informed consent provided by both parents for participation.
Sampling Method: Probability Sample
Enrollment: 111 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
KREC and CD19 of B-cells in offspring to mothers with MS exposed to monoclonal anti-CD20 antibodies | 2 years (2022-2023)
  Measurement of KREC and CD19 reflecting B-cells in offspring to women with MS who are exposed to monoclonal anti-CD20 antibodies before or during pregnancy compared to controls with MS and other DMT as well as MS without DMT.
Antibody production post vaccination in offspring to mothers with MS exposed to monoclonal anti-CD20 antibodies | 4 years (2022-2025)
  Measurement of antibody response to vaccination 1-12 months post vaccination in children of of mothers with MS exposed to anti-CD20 antibodies compared to control groups with other DMT and no DMT respectively.
Frequency and severity of infections in mothers with MS exposed to monoclonal anti-CD20 antibodies and their offspring | 4 years (2022-2025)
  Evaluation through history at clinical follow up and measurement of hypogammaglobulinemia in mother at every trimester and 3 months post partum as part of routine follow up.
Blood levels of monoclonal anti-CD20 antibodies in offspring to mothers with MS exposed to monoclonal anti-CD20 antibodies before or during pregnancy | 4 years (2022-2025)
  Measurement of anti-CD20 antibodies in dry blood spot from blood samples collected and stored at birth in offspring to mothers with MS
Levels of monoclonal anti-CD20 antibodies in breastmilk of breastfeeding mothers treated with monoclonal anti-CD20 antibodies in addition to measurement of anti-CD20 antibodies and evaluation of B-cells in blood from the breastfed child | 4 years (2022-2025)
  Mothers with MS exposed to monoclonal anti-CD20 antibodies who choose to breastfeed may transfer antibodies to their child. Measurements of monoclonal anti-CD20 antibodies as well as a potential effect on childs B-cells one month post treatment hold potential to clarify this.

CONTACTS AND LOCATIONS:
Overall Officials: Sofia Ernestam, MD, PhD, Study Director — Karolinska Institutet

IPD SHARING:
Plan to Share IPD: Yes
All IPD will be available in a Microsoft Excel file with encoded access to researchers participating in the study. IPD will be made anonymized through a coding system and non anonymized data will only be available when necessary e.g connection between CMMS and patients clinical notes. IPD will be shared anonymously according to below when study results are published according to routine scientific methods.Complete data set will be stored 10 years post publication in anonymous format.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 2025-2035
Access Criteria: Access to researchers who are part of the study project through approval from Dr Katharina Fink

REFERENCES:
- [Background] Ahlgren C, Oden A, Lycke J. High nationwide incidence of multiple sclerosis in Sweden. PLoS One. 2014 Sep 29;9(9):e108599. doi: 10.1371/journal.pone.0108599. eCollection 2014. PMID 25265372
- [Background] Bove R, Alwan S, Friedman JM, Hellwig K, Houtchens M, Koren G, Lu E, McElrath TF, Smyth P, Tremlett H, Sadovnick AD. Management of multiple sclerosis during pregnancy and the reproductive years: a systematic review. Obstet Gynecol. 2014 Dec;124(6):1157-1168. doi: 10.1097/AOG.0000000000000541. PMID 25415167
- [Background] Langer-Gould AM. Pregnancy and Family Planning in Multiple Sclerosis. Continuum (Minneap Minn). 2019 Jun;25(3):773-792. doi: 10.1212/CON.0000000000000745. PMID 31162316
- [Background] Stern J, Salih Joelsson L, Tyden T, Berglund A, Ekstrand M, Hegaard H, Aarts C, Rosenblad A, Larsson M, Kristiansson P. Is pregnancy planning associated with background characteristics and pregnancy-planning behavior? Acta Obstet Gynecol Scand. 2016 Feb;95(2):182-9. doi: 10.1111/aogs.12816. Epub 2015 Dec 8. PMID 26566076
- [Background] Sedgh G, Singh S, Hussain R. Intended and unintended pregnancies worldwide in 2012 and recent trends. Stud Fam Plann. 2014 Sep;45(3):301-14. doi: 10.1111/j.1728-4465.2014.00393.x. PMID 25207494
- [Background] Bearak J, Popinchalk A, Alkema L, Sedgh G. Global, regional, and subregional trends in unintended pregnancy and its outcomes from 1990 to 2014: estimates from a Bayesian hierarchical model. Lancet Glob Health. 2018 Apr;6(4):e380-e389. doi: 10.1016/S2214-109X(18)30029-9. Epub 2018 Mar 5. PMID 29519649
- [Background] Salzer J, Svenningsson R, Alping P, Novakova L, Bjorck A, Fink K, Islam-Jakobsson P, Malmestrom C, Axelsson M, Vagberg M, Sundstrom P, Lycke J, Piehl F, Svenningsson A. Rituximab in multiple sclerosis: A retrospective observational study on safety and efficacy. Neurology. 2016 Nov 15;87(20):2074-2081. doi: 10.1212/WNL.0000000000003331. Epub 2016 Oct 19. PMID 27760868
- [Background] Klink DT, van Elburg RM, Schreurs MW, van Well GT. Rituximab administration in third trimester of pregnancy suppresses neonatal B-cell development. Clin Dev Immunol. 2008;2008:271363. doi: 10.1155/2008/271363. PMID 18596903
- [Background] Kumpfel T, Thiel S, Meinl I, Ciplea AI, Bayas A, Hoffmann F, Hofstadt-van Oy U, Hoshi M, Kluge J, Ringelstein M, Aktas O, Stoppe M, Walter A, Weber MS, Ayzenberg I, Hellwig K. Anti-CD20 therapies and pregnancy in neuroimmunologic disorders: A cohort study from Germany. Neurol Neuroimmunol Neuroinflamm. 2020 Dec 17;8(1):e913. doi: 10.1212/NXI.0000000000000913. Print 2021 Jan. PMID 33334856
- [Background] Smith JB, Hellwig K, Fink K, Lyell DJ, Piehl F, Langer-Gould A. Rituximab, MS, and pregnancy. Neurol Neuroimmunol Neuroinflamm. 2020 May 1;7(4):e734. doi: 10.1212/NXI.0000000000000734. Print 2020 Jul. PMID 32358226
- [Background] Perrotta K, Kiernan E, Bandoli G, Manaster R, Chambers C. Pregnancy outcomes following maternal treatment with rituximab prior to or during pregnancy: a case series. Rheumatol Adv Pract. 2021 Jan 4;5(1):rkaa074. doi: 10.1093/rap/rkaa074. eCollection 2021. PMID 33521513
- [Background] Hollen C, Rice J, Park M, Yadav V. Rituximab for treatment of refractory multiple sclerosis relapses during pregnancy. Mult Scler. 2021 Sep;27(10):1620-1623. doi: 10.1177/1352458521998937. Epub 2021 Apr 30. PMID 33929267
- [Background] Routes JM, Grossman WJ, Verbsky J, Laessig RH, Hoffman GL, Brokopp CD, Baker MW. Statewide newborn screening for severe T-cell lymphopenia. JAMA. 2009 Dec 9;302(22):2465-70. doi: 10.1001/jama.2009.1806. PMID 19996402
- [Background] Borte S, von Dobeln U, Fasth A, Wang N, Janzi M, Winiarski J, Sack U, Pan-Hammarstrom Q, Borte M, Hammarstrom L. Neonatal screening for severe primary immunodeficiency diseases using high-throughput triplex real-time PCR. Blood. 2012 Mar 15;119(11):2552-5. doi: 10.1182/blood-2011-08-371021. Epub 2011 Nov 30. PMID 22130802
- [Background] Schrezenmeier E, Jayne D, Dorner T. Targeting B Cells and Plasma Cells in Glomerular Diseases: Translational Perspectives. J Am Soc Nephrol. 2018 Mar;29(3):741-758. doi: 10.1681/ASN.2017040367. Epub 2018 Jan 11. PMID 29326157
- [Background] Kruger R, Borte S, von Weizsacker K, Wahn V, Feiterna-Sperling C. Positive Kappa-Deleting Recombination Excision Circles (KREC) Newborn Screening in a Neonate With Intrauterine Exposure to Rituximab. Scand J Immunol. 2018 Jan;87(1):54-56. doi: 10.1111/sji.12627. No abstract available. PMID 29106704
- [Background] Barbaro M, Ohlsson A, Borte S, Jonsson S, Zetterstrom RH, King J, Winiarski J, von Dobeln U, Hammarstrom L. Newborn Screening for Severe Primary Immunodeficiency Diseases in Sweden-a 2-Year Pilot TREC and KREC Screening Study. J Clin Immunol. 2017 Jan;37(1):51-60. doi: 10.1007/s10875-016-0347-5. Epub 2016 Nov 21. PMID 27873105
- [Background] Serana F, Chiarini M, Zanotti C, Sottini A, Bertoli D, Bosio A, Caimi L, Imberti L. Use of V(D)J recombination excision circles to identify T- and B-cell defects and to monitor the treatment in primary and acquired immunodeficiencies. J Transl Med. 2013 May 9;11:119. doi: 10.1186/1479-5876-11-119. PMID 23656963